CLINICAL TRIAL: NCT05925920
Title: A First in Human, Single Center, Single Dose, Randomized, Placebo-controlled, Dose, Escalating Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Subcutaneously Administered ENT-03S for the Treatment of Obesity and Diabetes
Brief Title: Study of Subcutaneously Administered ENT-03 for the Treatment of Obesity and Diabetes
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Metabolics Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: ENT-03S-22-001
Record Dates: First submitted 2023-06-05; First posted 2023-06-29 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Obesity; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Receive a single dose of ENT-03 sub-cutaneously
  Interventions: Drug: ENT-03
- Placebo (Placebo Comparator): Receive a single dose of placebo sub-cutaneously
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ENT-03 — single dose of active drug
  Arms: Active
Drug: Placebo — single dose of placebo comparator
  Arms: Placebo

SUMMARY:
Single center, single-dose, randomized, placebo-controlled, dose-escalating study to evaluate, safety, tolerability, pharmacokinetics, and pharmacodynamics of escalating doses of ENT-03S in obese but otherwise healthy subjects and in subjects with obesity and Type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18-70 years, both genders.
2. Healthy as determined by a physician, based on history, medical examination, vital signs, and laboratory tests.
3. Males that agree to use condoms for the duration of participation in the study.
4. Females of non-child-bearing potential (i.e., tubal ligation, hysterectomy, or postmenopausal).
5. Female patients of child-bearing potential with negative serum pregnancy tests and who agree to use double-barrier contraception during the study.
6. Subjects must be able to read, speak, and understand English and/or Spanish and provide written informed consent, and be willing and able to comply with study procedures.
7. Subjects must have a BMI 30-35 kg/m2 inclusive assessed immediately prior to screening.
8. Fasting insulin level ≥11 mIU/L.
9. HbA1c < 8.5% (diabetic subjects only).
10. Subjects with Type 2 diabetes on no anti-diabetic medication or on stable doses of metformin for 4 weeks or more (diabetic cohorts only).
11. No history of active or chronic disease other than that allowed by study: hypertension, hyperlipidemia, hyperglycemia, GERD, heartburn, or Type 2 diabetes (cohorts 6 and 7 only).

Exclusion Criteria:

1. History of excessive alcohol use (defined as >21 drinks per week for males and >14 drinks per week for females), recreational drug use within the past three months, or failure on urinary drug screen.
2. Pregnant or breastfeeding within six months of screening assessment.
3. Substantial changes in eating habits or exercise routine within the preceding three months.
4. Evidence of eating disorders.
5. >5% weight change in the past three months.
6. Bariatric surgery within the past five years.
7. Significant renal impairment (eGFR <60 mg/mL/1.73m2).
8. Patients on anti-diabetic medications other than metformin.
9. Patients with gastroparesis.
10. Liver function tests (i.e., ALT, AST, alkaline phosphatase) greater than twice the upper limit of normal upon repeated measurements.
11. Diseases interfering with metabolism and/or ingestive behavior (e.g., myxedema, Cushing's disease, schizophrenia, major psychoses).
12. History of major depressive disorder within the previous two years, a lifetime history of suicide attempt, suicidal behavior within the previous month, or history of other severe psychiatric disorders.
13. Score of >15 on the Columbia Suicide Severity Rating Scale (C-SSRS).
14. Use of medications affecting body weight within the past three months:

    * Drugs approved for the treatment of obesity
    * Cyproheptadine or medroxyprogesterone
    * Atypical anti-psychotic drugs
    * Tricyclic antidepressants
    * Lithium, MAO's, glucocorticoids
    * SSRI's or SNRI's
    * Antiepileptic drugs
15. Any clinically significant abnormality following the Investigator's review of the physical examination and clinical laboratory tests.
16. A baseline prolongation of QT/QTc interval after repeated measurements of >450 ms; a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsades de pointes, structural heart disease, or a family history of Long QT Syndrome (LQTS).
17. Participation in an investigational drug trial within the month prior to dosing in the present study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-12-06 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of ENT-03 | 7 days
  Adverse Events
Safety and Tolerability of ENT-03 | 7 days
  ECG: QTc analysis
Safety and Tolerability of ENT-03 | 7 days
  Vital signs: body temperature
Safety and Tolerability of ENT-03 | 7 days
  Vital signs: respiration rate
Safety and Tolerability of ENT-03 | 7 days
  Vital signs: heart rate
Safety and Tolerability of ENT-03 | 7 days
  Vital signs: systolic blood pressure measurements
Safety and Tolerability of ENT-03 | 7 days
  Vital signs: diastolic blood pressure measurements
Safety and Tolerability of ENT-03 | 7 days
  Vital signs: body weight in kilograms

SECONDARY OUTCOMES:
pharmacokinetic endpoints: maximum plasma concentration | pre-dose, 24 hours, 48 house, 72 hours
  maximum measured plasma concentration
pharmacokinetic endpoints: time of maximum plasma concentration | pre-dose, 24 hours, 48 house, 72 hours
  time of maximum measured plasma concentration
pharmacokinetic endpoints: ENT-03 half-life | pre-dose, 24 hours, 48 house, 72 hours
  terminal elimination of ENT-03 half-life in plasma
pharmacokinetic endpoints: plasma concentration | pre-dose, 24 hours, 48 house, 72 hours
  area under the concentration versus time curve over 24 hours
pharmacokinetic endpoint: ENT-03 clearance | pre-dose, 24 hours, 48 house, 72 hours
  Clearance of ENT-03
pharmacokinetic endpoint: elimination phase | pre-dose, 24 hours, 48 house, 72 hours
  slope of terminal elimination phase
pharmacodynamic endpoint: glucose | 7 days
  change from screening visit in fasting plasma glucose
pharmacodynamic endpoint: insulin | 7 days
  change from screening visit in fasting serum insulin
pharmacodynamic endpoint: fasting lipids | 7 days
  change from screening visit in fasting lipids
pharmacodynamic endpoint: fasting leptin | 7 days
  change from screening visit in fasting leptin
pharmacodynamic endpoint: body weight | 7 days
  change from screening visit in body weight (kg)
effect on glucose | Days -7, 2, 3, 4, and 7
  results of fasting and post-prandial blood glucose in subjects with obesity and T2D
effect on insulin and insulin sensitivity | Days -7, 2, 3, 4, and 7
  results of fasting and post-prandial blood insulin and insulin sensitivity as measured by homeostatic assessment of insulin resistance (HOMAIR), in subjects with obesity and T2D

CONTACTS AND LOCATIONS:
Overall Officials: Richard Larson, MD, Study Director — Enterin Inc.
Locations (1):
- ProSciento, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No